CLINICAL TRIAL: NCT05707065
Title: Comparative Effects of Core Strengthening Versus Lower Limb Proprioceptive Neuromuscular Facilitation Techniques on Trunk Function and Balance in Chronic Stroke Patients
Brief Title: Core Strengthening Versus Lower Limb Proprioceptive Neuromuscular Facilitation Techniques in Chronic Stroke Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/22/0217
Record Dates: First submitted 2023-01-22; First posted 2023-01-31 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Stroke
Keywords: Proprioceptive Neuromuscular Facilitation; Stroke
MeSH Terms: conditions — Stroke | interventions — Muscle Stretching Exercises

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- core strengthening exercises (Experimental): Participants will be positioned in supine.
  * first stage participants will be taught to activate abdominal wall musculature. They will be initially trained to perform abdominal bracing.
  * Then positioned in quadruped position and asked to lift alternate arms, gradually progressing to alternate leg lifts and alternate arm/leg raises to activate multifidus.
  * Then side bridges (side plank) exercise for activation of quadratus lumborum and obliques.
  * Then asked to perform trunk curls in crook lying, asking them to lift their upper trunk slightly (15°) from the plinth, hold the position for 5 sec.
  * Perform 30 repetitions of each exercise with 8-sec hold.
  * Maintain normal diaphragmatic breathing throughout the intervention
  Interventions: Other: core strengthening exercises
- Proprioceptive Neuromuscular Facilitation (Experimental): * Rhythmic initiation (RI) Patients progressively performed voluntary relaxation, passive movements, active assisted, active resisted movements and than active movements.
  * Dynamic reversals (slow reversals) Isotonic contractions of first agonists and then antagonists performed against resistance was performed initially.
  * Stabilizing reversals Isotonic contractions of first agonists, then antagonists against resistance was performed in an alternate way.
  * Mixture of isotonic (agonist reversals, AR) resisted concentric, contraction of agonist muscles moving with the range was performed progressively following eccentric, lengthening contraction, moving slowing to the start position. .
  Total 30 min for 3 days a week for a total duration of 4 weeks was set as a optimal time frame duration. Each technique was given for 10 min.
  Interventions: Other: Proprioceptive Neuromuscular Facilitation

INTERVENTIONS:
Other: core strengthening exercises — The core muscles training includes transverse abdominis, multifidus, paraspinals, quadratus lumborum, and obliques.
  Arms: core strengthening exercises
Other: Proprioceptive Neuromuscular Facilitation — lower limb PNF technique along with conventional treatment i.e., Rhythmic initiation, slow reversal, stabilizing reversal, and combination of isotones.
  Arms: Proprioceptive Neuromuscular Facilitation

SUMMARY:
Stroke is a global healthcare issue that causes increased death rates. Good trunk stability is essential for balance and extremity use during daily functional activities and higher-level tasks. The anticipatory activity of trunk muscles is impaired in stroke patients. The trunk is the central column of the body; therefore, proximal trunk control is a prerequisite for distal limb movement control, balance, and functional activities. The purpose of the study is to highlight the most appropriate rehabilitation technique for trunk stability.

DETAILED DESCRIPTION:
A randomized clinical trial will be performed in which 42 patients with strokes will be included. The data will be collected from Riphah Rehabilitation center Lahore and Ittefaq hospital Lahore. Consecutive sampling technique will be used to collect data. The duration of the study will be 10 months. Trunk impairment scale and berg balance scale will be used as the data collection tool. Data collection will be started after taking informed consent from all the patients. Patients will be allocated to intervention groups by randomization. The patients in group A will be given core strengthening exercise for 4 weeks. The patient in group B will be given PNF exercise for the treatment of trunk for 4 weeks. After data collection analysis of pre and post values will be done by using SPSS version 25.

ELIGIBILITY:
Inclusion Criteria:

* Chronic stroke patients (6 months to 2 years).
* Participants with first ever ischemic stroke of right or left half of the body.
* Participants should be able to walk without support for 10 m.
* MMSE score is ≥ 24.

Exclusion Criteria:

* Participants with recurrent stroke; brainstem or cerebellar stroke or hemorrhagic stroke will be excluded.
* Patients with speech problem after stroke
* Patients with other neurological disorders including: Parkinson's disease, multiple sclerosis, epilepsy, etc.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-03-15 (Estimated); Study Completion 2023-03-22 (Estimated)

PRIMARY OUTCOMES:
Berg balance scale | 4th week
  Changes from baseline Berg balance scale is used to objectively determine a patient's ability (or inability) to safely balance during a series of predetermined tasks. It is a 14-item list with each item consisting of a five-point ordinal scale ranging from 0 to 4, with 0 indicating the lowest level of function and 4 the highest level of function and takes approximately 20 minutes to complete. It does not include the assessment of gait.
Trunk Impairment Scale (TIS) | 4th week
  Changes from baseline TIS is a new tool to measure motor impairment of the trunk after stroke. The TIS evaluates static and dynamic sitting balance as well as co-ordination of trunk movement.

CONTACTS AND LOCATIONS:
Overall Officials: Ali Raza, MS(OMPT), Principal Investigator — Riphah International University
Locations (1):
- Ittefaq Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sharma V, Kaur J. Effect of core strengthening with pelvic proprioceptive neuromuscular facilitation on trunk, balance, gait, and function in chronic stroke. J Exerc Rehabil. 2017 Apr 30;13(2):200-205. doi: 10.12965/jer.1734892.446. eCollection 2017 Apr. PMID 28503533
- [Background] Park SE, Moon SH. Effects of trunk stability exercise using proprioceptive neuromuscular facilitation with changes in chair height on the gait of patients who had a stroke. J Phys Ther Sci. 2016 Jul;28(7):2014-8. doi: 10.1589/jpts.28.2014. Epub 2016 Jul 29. PMID 27512254
- [Background] Suh JH, Lee EC, Kim JS, Yoon SY. Association between trunk core muscle thickness and functional ability in subacute hemiplegic stroke patients: an exploratory cross-sectional study. Top Stroke Rehabil. 2022 Apr;29(3):163-172. doi: 10.1080/10749357.2021.1918840. Epub 2021 Apr 26. PMID 33899701
- [Background] Asghar M, Fatima A, Warner S, Khan MHU, Ahmad A, Siddique K. Effectiveness of proprioceptive neuromuscular facilitation on balance in chronic stroke patients. Rawal Medical Journal. 2021;46(1):212-5
- [Background] Krukowska J, Bugajski M, Sienkiewicz M, Czernicki J. The influence of NDT-Bobath and PNF methods on the field support and total path length measure foot pressure (COP) in patients after stroke. Neurol Neurochir Pol. 2016 Nov-Dec;50(6):449-454. doi: 10.1016/j.pjnns.2016.08.004. Epub 2016 Aug 20. PMID 27585746